CLINICAL TRIAL: NCT05396664
Title: Adolescent Transition West Africa: An Outcome Evaluation of a Gender and Sexual and Reproductive Health and Rights Intervention in Mali, Burkina Faso, and Niger
Brief Title: Adolescent Transition West Africa
Acronym: ATWA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Save the Children Netherlands (Unknown); GRADE Africa (Unknown)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111111
Record Dates: First submitted 2022-01-19; First posted 2022-05-31 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Adolescent Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ATWA LSE program will be implemented following a joint curricula development process with approval from the government in each of the three countries. The 'dose' of the intervention are once-weekly hour-long sessions for both in-school adolescents (session facilitated by teachers) and out-of-school adolescents (sessions facilitated by community leaders) over the course of the academic year (roughly 9 months), or roughly 30 sessions of exposure to the in-depth LSE curriculum.
  Interventions: Behavioral: ATWA
- Control (No Intervention): Control groups are comprised of adolescents (10-19) attending schools where the ATWA Life Skills Education (LSE) program has not been implemented, as well as out-of-school adolescents (10-19) who have not received the ATWA LSE program in their communities. Control groups receive "standard of care" educational opportunities. "Standard of care" in the case of this trial translate to the provision of standard Ministry of Education-sanctioned sexuality education, as already available in the adolescents' schools and communities.

INTERVENTIONS:
Behavioral: ATWA — The Adolescent Transition in West Africa (ATWA) program is an in-school (Niger, Mali, Burkina Faso) and out-of-school (Niger and Mali) educational intervention implemented by local staff members at Save the Children, local community members, and teachers. ATWA provides internationally-recognized life skills education (LSE) to adolescents ages 10-19 years, and seeks to improve adolescents' knowledge and behaviors regarding sexual and reproductive health and rights. Outcome indicators to assess knowledge, behavior and attitudes of adolescents will vary by adolescent demographics as well as by country context, as based on the final set of curriculum deemed appropriate by the respective Ministries of Education (MOE).
  Arms: Intervention

SUMMARY:
This trial will serve as an outcome evaluation of 'Adolescent Transition in West Africa' (ATWA), a school-based program in Mali, Burkina Faso, and Niger for adolescents ages 10-19. The overall objectives of the project are as follows: Impact: Improved sexual and reproductive health and rights of 472,180 adolescents. Outcome 1: Improved sexual and reproductive health and rights and gender equality knowledge, intent, and behaviors among 472,180 adolescents. Outcome 2: 500 health facilities offer quality adolescent responsive SRH services that are used by adolescent girls and boys. To evaluate program impact, an external evaluation will be conducted. A pre/post cross-sectional evaluation design will be used across two evaluation years.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in primary or secondary school
* Participating in community group (Niger only)
* Aged 10 to 19

Exclusion Criteria:

* Not enrolled in school (Mali and Burkina Faso)
* Younger than age 10
* Older than age 19

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4300 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Impact Indicator 1. Decrease in adolescent birth rate | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  The average number of births to female respondents ages 15-19
Impact 2. Decrease in proportion of adolescents who have ever been pregnant or caused a pregnancy | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  The percent of adolescent females who have ever been pregnant + the percent of adolescent males who have ever caused a pregnancy
Impact 3. Increase in need for family planning satisfied with modern contraception | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Indicator definition 3A: Percentage of [sexually active] adolescents age 15-19 years currently married or in union who have their need for family planning satisfied with modern contraceptive methods Indicator definition 3B: Percentage of female adolescents (15-19) who are sexually active and who have their need for contraception satisfied with modern methods
Impact 4. Increase in adolescent modern contraceptive prevalence rate | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  The percent of sexually active adolescents (15-19) who are currently using (or whose partner is using) a modern contraceptive method. "Currently" is defined as 'at last sex'
Impact 5. Decrease in proportion of adolescents married | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Indicator definition 5A: Percentage of women 10-19 years old living with spouse before age 18.
  Indicator definition 5B: Percentage of women 10-19 years old living with spouse before age 15.
Outcome 1.1. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents who respond yes to planning to use modern contraception in the future, disaggregated by method
Outcome 1.2. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of sexually active adolescents reporting using a condom at last sex
Outcome 1.3. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of sexually active unmarried adolescents who respond yes to having used a condom every time they had sex in the last 6 months
Outcome 1.4. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents with significant increase from baseline to end-line in average score on a 6-item gender equitable attitude scale
Outcome 1.5. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Average number of modern contraceptive methods known among women 10-14 and 15-19 years old
Outcome 1.6. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents with correct knowledge about body changes during puberty, the menstrual cycle, fertility and conception, pregnancy risk and prevention, as assessed via a 9-item composite indicator
Outcome 1.7. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents with correct knowledge about STI risk and prevention and treatment, assessed using a composite indicator of 4 questions on STI prevention and treatment
Outcome 1.8. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents with comprehensive knowledge of HIV prevention, assessed using a composite indicator of 6 questions on HIV prevention
Outcome 1.9. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of adolescents with knowledge of where to seek SRH services, including where to get tested for HIV, where to get condoms, and where to get contraceptives
Outcome 1.10. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of girls who report properly disposing of absorbent materials (sanitary napkins or menstrual cloth) (denominator = the total number of girls who use absorbent materials (sanitary napkins or menstrual cloth))
Outcome 1.11. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of girls who report hygienically washing and drying reusable menstrual cloth (denominator = number of girls who washed and reused menstrual materials)
Output 1.2.1. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of girls and boys that can correctly answer a basic set of four yes/no questions about menstruation
Output 1.2.2. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of girls that can answer a set of five questions correctly about how to hygienically manage menses
Output 1.2.3. | Year 1 Evaluation: September 2021 - May 2022; Year 2 Evaluation: September 2022 - May 2023
  Proportion of girls and boys that answer a question correctly regarding that menstruation is a normal biological function of the female body

CONTACTS AND LOCATIONS:
Overall Officials: Jay Silverman, PhD, Principal Investigator — University of California, San Diego
Locations (3):
- Save the Children, Burkina Faso, Ouagadougou, Burkina Faso
- Save the Children, Mali, Bamako, Mali
- Save the Children, Niger, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No